CLINICAL TRIAL: NCT01568905
Title: Palatability of Experimental Cigarettes
Brief Title: Palatability of Experimental Cigarettes - Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 1012M94314
Record Dates: First submitted 2012-01-03; First posted 2012-04-02 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Smoking
Keywords: smoker; smoking; nicotine levels; tobacco; nicotine
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 Low Level Nicotine Cigarette (Experimental): (0.4 mg/g)
  Interventions: Other: Low level nicotine cigarette
- Arm 2 Intermediate Nicotine Level Cigarette (Experimental): (5.7-5.8 mg/g)
  Interventions: Other: Intermediate nicotine level cigarette
- Arm 3 High Level Nicotine Cigarette (Experimental): (11.4-12.8 mg/g)
  Interventions: Other: High level nicotine cigarette

INTERVENTIONS:
Other: Low level nicotine cigarette — smoke the study cigarette exclusively for one week
  Arms: Arm 1 Low Level Nicotine Cigarette
Other: Intermediate nicotine level cigarette — smoke the study cigarette exclusively for one week
  Arms: Arm 2 Intermediate Nicotine Level Cigarette
Other: High level nicotine cigarette — smoke the study cigarette exclusively for one week
  Arms: Arm 3 High Level Nicotine Cigarette

SUMMARY:
Smoking remains a leading cause of preventable disease and premature death worldwide. Approximately 1 out of every 5 deaths is associated with cigarette smoking, and roughly half of all daily smokers will die prematurely from tobacco-related illness. Reducing the nicotine in cigarettes to the point that they are rendered non-addictive can potentially be an effective public policy measure that can significantly reduce tobacco-related mortality and morbidity by decreasing the initiation of smoking and promoting cessation. The Family Smoking Prevention and Tobacco Control Act (FSPTCA) enables the FDA to establish tobacco product standards including placing limits on the allowable nicotine content of cigarettes. Currently, no reduced nicotine cigarettes are available that will allow studying the feasibility of this policy measure. The National Institute on Drug Abuse has contracted with Research Triangle Institute to assist in the development of cigarettes with varying nicotine content that can be made available to researchers. They have established a contract that will result in the manufacture of 9 million cigarettes to be distributed to the research community. Prior to full production, the palatability and nicotine intake of these cigarettes in smokers must be determined.

DETAILED DESCRIPTION:
Phase 3: This descriptive study will use a between subjects, double blind design. This study will test 3 nicotine levels of nicotine, tar and ventilation. Subjects and research assistants will be blind to the cigarette type.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old
* Regular smokers (10+ cigarettes per day and has done so for the last year)
* Inhaling when smoking
* Carbon monoxide (CO) > 8 ppm

Exclusion Criteria:

* In the past year, suffered from any cardiovascular disease such as: heart disease, heart attack, stroke or angina, any respiratory diseases such as chronic bronchitis or chronic obstructive pulmonary disease (COPD), any type of cancer
* Currently suffering from Bipolar Disorder, General Anxiety Disorder, Schizophrenia, or a major depressive episode
* Taken any of the following drugs more than twice per week during the past month: antidepressants, anti-anxiety medications.
* Consumed more than 15 alcoholic drinks per week for the past month
* Pregnant, trying to become pregnant, or lactating (assessed by self-report)
* In the past 3 months, used nicotine replacement products (like the patch, gum, or inhaler), or the medications bupropion varenicline
* Currently trying or planning to reduce or quit tobacco use in the next 30 days
* Used other forms of tobacco 10 or more days in the past 30 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, Ph.D., Principal Investigator — Tobacco Use Research Program, University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Hatsukami DK, Heishman SJ, Vogel RI, Denlinger RL, Roper-Batker AN, Mackowick KM, Jensen J, Murphy SE, Thomas BF, Donny E. Dose-response effects of spectrum research cigarettes. Nicotine Tob Res. 2013 Jun;15(6):1113-21. doi: 10.1093/ntr/nts247. Epub 2012 Nov 22. PMID 23178320

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Started | 13 | 11 | 12
Completed | 12 | 11 | 12
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Daily cigarette smokers
Groups:
- Arm 1 Low Level Nicotine Cigarette: Low level nicotine cigarette (0.400 mg/g; menthol 0.405 mg/g): smoke the study cigarette exclusively for one week
- Arm 2 Intermediate Nicotine Level Cigarette: Intermediate nicotine level cigarette (5.86 mg/g menthol 5.87 mg/g): smoke the study cigarette exclusively for one week
- Arm 3 High Level Nicotine Cigarette: High level nicotine cigarette (10.4 mg/g; menthol: 12.3): smoke the study cigarette exclusively for one week
- Total: Total of all reporting groups
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette | Total
Number analyzed (Participants) | 12 | 11 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 12 | 35
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.4) | 32.7 (10.8) | 43.6 (9.6) | 37.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 5 | 20
  Male | 4 | 4 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 12 | 35
Menthol [Number; unit: participants]
  Menthol | 4 | 3 | 4 | 11
  Non Menthol | 8 | 8 | 8 | 24
Cigarettes per day [Mean (Standard Deviation); unit: Cigarettes per day] | 16.8 (5.1) | 16.1 (3.5) | 18.7 (4.3) | 17.2 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in UrineTotal Nicotine Equivalent (TNE) Between Baseline and Week 1
Description: Two urine TNE levels are taken, one at baseline and one at week 1, to assess TNE levels for nicotine exposure. TNE is the sum of nicotine, cotinine, trans 3'-hydroxycotinine and their respective glucuronide conjugates. Values reported in nmols/ml.
Time Frame: Second Visit (Week 1) minus Baseline (Day 1)
Measure: Mean (Standard Error); unit: nmols/ml
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Number analyzed (Participants) | 12 | 11 | 12
nmols/ml | -16.2 (5.0) | -7.6 (4.7) | 1.3 (4.4)

2. Secondary Outcome: Responses on Modified Cigarette Evaluation Scale
Description: Modified Cigarette Evaluation Scale [CES] is a 100 mm visual analog scale (0=not at all or very little nicotine; 100=extremely or high in nicotine) of 20 questions assessing different dimensions of responses to usual brand cigarettes (e.g., psychological reward, satisfaction and aversiveness) and includes additional 5 point likert-type questions (definitely agree to definitely disagree) on perceptions of satisfaction and willingness to use the product. Results satisfaction subscale.
Time Frame: Baseline usual brand cigarettes (Day 1) compared to when using study cigarettes (Week 1)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Number analyzed (Participants) | 12 | 11 | 12
units on a scale | 36.8 (4.1) | 54.1 (4.1) | 61.4 (4.1)

3. Secondary Outcome: Change From Baseline of Perceived Health Risk Scale Response to Test Cigarettes
Description: Questionnaire: Perceived Health Risk Scale asks subjects to rate their perception of health risks for lung cancer for the study product to which they have been randomly assigned. This is a 100 mm visual analog scale; 0=very low risk of disease, 100=very high risk of disease.
Time Frame: Baseline (Day 1) Compared to Second Visit (Week 1)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Number analyzed (Participants) | 12 | 11 | 12
units on a scale | 56.6 (4.6) | 66.7 (4.6) | 68.3 (4.6)

4. Secondary Outcome: Comparison of Number of Cigarettes Smoked
Description: Subjects were given a daily diary to collect the number of study and/or conventional cigarettes they have smoked each day. Cigarettes smoked (both usual brand and experimental) in a given week were summed over the first 7 reported days. If the number of cigarettes smoked was missing for 1 day, the average of the other days in that week was used in its place and reported as total number of cigarettes per week.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: cigarettes per week
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Number analyzed (Participants) | 12 | 11 | 12
cigarettes per week | 92.1 (15.9) | 112.8 (49.4) | 157.6 (15.2)

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Arm 1 Low Level Nicotine Cigarette | Arm 2 Intermediate Nicotine Level Cigarette | Arm 3 High Level Nicotine Cigarette
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No